CLINICAL TRIAL: NCT02422043
Title: Description of Socio-cognitive and Clinic Changes for Type 1 Diabetes Adolescents Cohort With Therapeutic Patient Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-28
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Type 1 Diabetes
Keywords: adolescence
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- type 1 diabetes adolescents cohort (Experimental): The participants of the prospective cohort of adolescents will be 12 to 17 years of age, type 1 diabetics with insulin, included in TPE program
  Interventions: Other: Questionnaires and audio-tape interviews

INTERVENTIONS:
Other: Questionnaires and audio-tape interviews — therapeutic patient education programs (TPE) to type 1 diabetic adolescents are designed to make the teenager to self manage their disease and their treatment. Based on Bandura's social cognitive theory, effects of educational activities for TPE should lead to the strengthening of self-efficacy

SUMMARY:
The patient education programs (TPEs) for the type 1 diabetic adolescents are designed to make the teenager to self manage their disease and its treatment. Based on social cognitive theory Bandura, the effects of educational activities for TVE should lead to the strengthening of self-efficacy, coupled with other socio-cognitive factors favoring adherence of teenager and a better quality of life. However, socio-cognitive determinants and mechanisms to achieve this, implemented by adolescents during and after the ETP program, are not sufficiently documented.

DETAILED DESCRIPTION:
Therapeutic patient education programs (TPE) to type 1 diabetic adolescents are designed to make the teenager to self manage their disease and their treatment. Based on Bandura's social cognitive theory, effects of educational activities for TPE should lead to the strengthening of self-efficacy, coupled with other socio-cognitive factors favoring adherence and a better quality of life for teenager. However, socio-cognitive determinants and mechanisms to achieve this, implemented by adolescents during and after the TPE program, are not sufficiently documented and French assessment tools are missing.

Objectives: The main objective of the research is to validate self-efficacy and adherence tools in French for type 1 diabetic teenagers, and secondarily, to describe evolution of a 3-month cohort of type 1 diabetes adolescents who took a TPE program on self-efficacy, quality of life, adherence, glycated hemoglobin (HbA1c) and socio-cognitive factors as Bandura's social cognitive theory and the study of possible links between these endpoints.

The participants of the prospective cohort of adolescents will be 12 to 17 years of age, type 1 diabetics with insulin, included in TPE program in one of two study areas. The number of subjects required was estimated to 80 patients. The process of cross-cultural adaptation tools will be through a linguistic and metrological validation. An integrated mixed method was used, consisting of three components:

* A quantitative before-after study: Collection and analysis of changes over 3 months of self-efficacy, adherence, quality of life and HbA1c (Student t test);
* A longitudinal qualitative study: interviews with 24 participants M0, M1 and M3 on the socio-cognitive factors according to Bandura (analysis continues theming)
* An integrative component: exploratory data analysis methods in order to link the evolution of treatment adherence and quality of life, with the evolution of self-efficacy and additional socio-cognitive factors.

Outcomes: This pilot research should validate the assessment tools and improve educational sessions for existing and future TPE programs, to type 1 diabetic teenagers to enhance their particular self-efficacy and to promote their independence and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Aged between 12 and 17 inclusive; Type 1 diabetes diagnosis confirmed by a physician according to the diagnostic criteria (IDF & ISPAD, 2011); Length of more than 6 months in the disease; Treatment with insulin for at least 6 months before the educational intervention; Inclusion in a TPE program "Pediatric Diabetes" allowed by the Regional Health Agency Mastery of the French language in written form (elementary level); Mastery of speaking the French language (elementary level); Consent signed by the holders of parental authority and adolescents.

Exclusion Criteria:

Adolescents considered treatment failure, addressed to the SSR for intensive TPE inpatient program over a period of more than a month; Pregnant women, breast-feeding mothers (art L.1121-5 CSP). Persons deprived of their liberty by a judicial or administrative decision, those hospitalized without consent under Articles L. 3212-1 and L. 3213-1 which do not fall under the provisions of Article L. 1121-8 and persons admitted to a health or social establishment for purposes other than research (art. L.1121-6 CSP) Major persons under a legal protection measure or unable to consent (Article L.1121-8 CSP).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
self-efficacy (Self-efficacy of Diabetes Management) | 3 months
  a10-items tools self-passation at M0-J2-M1 and M3

SECONDARY OUTCOMES:
Quality of life (KIDSCREEN-27) | 3 months
  a 27-items tools self-passation at M0-M1 and M3
Adherence (Diabetes Self-Management Profile) | 3 months
  a 35-items tools, completed during interview with health professional at M0-J2-M1 and M3
glycated hemoglobin (HbA1c) | 3 months
  Description: biological at M0 and M3
socio-cognitive profile | 3 months
  interviews at M0-M1 and M3

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France